CLINICAL TRIAL: NCT01398462
Title: A Phase I Clinical Study of CWP232291 in Patients With Relapsed or Refractory Acute Myeloid Leukemia or Chronic Myelomonocytic Leukemia-2, Myelodysplastic Syndrome Having Failed Hypomethylating Treatment, and High-Risk Myelofibrosis
Brief Title: Phase I Clinical Study of CWP232291 in Acute Myeloid Leukemia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JW-231A-101
Record Dates: First submitted 2011-07-17; First posted 2011-07-20 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome; Myelofibrosis
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CWP232291 (Experimental)
  Interventions: Drug: CWP232291

INTERVENTIONS:
Drug: CWP232291 — IV Infusion

SUMMARY:
CWP232291 blocks proliferation of cancer cells via activation of caspases. Active caspase have been shown to target beta-catenin, the hallmark of canonical Wnt signaling, for degradation through caspase-directed cleavage. CWP232291 targets beta-catenin for degradation and thereby inhibits the expression of cell cycle and anti-apoptotic genes such as cyclin D1 and survivin.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to sign an informed consent form (ICF) prior to initiation of any study-specific procedure and treatment
* 18 years of age
* 3. A pathologically confirmed diagnosis of AML or CMML-2 by World Health Organization (WHO) classification that is relapsed or refractory or for which no current therapies are anticipated to result in a durable remission, or MDS by WHO classification are RAEB-1 or RAEB-2 and that have failed at least three cycles of hypomethylating therapy, or primary (PMF), post-polycythemia vera (PPMF) or post-essential thrombocythemia (PTMF) MF by WHO classification, are high-risk category by the Dynamic International Prognostic Scoring System (DIPSS Plus), have ≥1% circulating blasts, and have failed treatment with ruxolitinib
* Eastern Cooperative Oncology Group (ECOG) performance score 0-2
* In the absence of rapidly progressing disease, the interval from prior treatment to time of study drug administration should be at least 2 weeks for cytotoxic agents or at least 5 half-lives for noncytotoxic agents. If a patient is on hydroxyurea to control peripheral blood leukemic cell counts, the patient must have discontinued hydroxyurea for at least 24 hours before initiation of treatment with study drug. Persistent clinically significant toxicities from prior chemotherapy must not be greater than grade 1
* Adequate renal function:

  * Serum creatinine =/< 2.0mg/dL
* Adequate hepatic function:

  * Total bilirubin <1.5 x upper limit of normal (ULN), unless considered due to Gilbert's syndrome
  * Alkaline phosphatase (AP) =/< 2.5 x ULN
  * Aspartate transaminase (AST) or alanine transaminase (ALT) ≤3 x ULN, unless considered due to organ leukemic involvement
* Women of child-bearing potential (i.e., women who are pre menopausal or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive, or double barrier device), and must have a negative serum or urine pregnancy test within 2 weeks prior to beginning treatment on this trial. Sexually active men must also use acceptable contraceptive methods for the duration of time on study
* Able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure (CHF), cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements
* Active heart disease including myocardial infarction (MI) within previous 3 months, symptomatic coronary artery disease (CAD), arrhythmias not controlled by medication, or uncontrolled CHF
* Active central nervous system (CNS) disease
* Therapy with any other standard or investigational treatment for hematologic malignancy (except hydroxyurea, as mentioned in the inclusion criteria)
* Therapy with anticoagulant or antithrombotic agents (including aspirin) within 7 days prior to study drug administration
* History of gastrointestinal (GI) hemorrhage
* Known positive status for human immunodeficiency virus (HIV) and/or active hepatitis B or C
* Pregnant or nursing women. Pregnant and nursing patients are excluded because the effects of CWP232291 on a fetus or nursing child are unknown.
* Patients eligible for bone marrow transplant, regardless of age
* Patients with FLT3 ITD positive AML or AML patients with other cytogenetic abnormalities who are eligible for trials of other targeted investigational agents from which the investigator feels there is greater benefit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Up to 3 weeks after start of injection
  If myelosuppression is DLT (Dose-Limiting Toxicity), it will be monitored up to 42 days after start of injection.

SECONDARY OUTCOMES:
Cmax as a pharmacokinetic parameter of 'CWP232291' | 0, 0.25, 0.5, 1, 1.5, 2, 4, 8, 24 hours post-dose
  Peak Plasma Concentration (Cmax) of 'CWP232291'
AUC as a pharmacokinetic parameter of 'CWP232291' | 0, 0.25, 0.5, 1, 1.5, 2, 4, 8, 24 hours post-dose
  Area under the plasma concentration versus time curve (AUC) of 'CWP232291'
Cmax as a pharmacokinetic parameter of metabolites of 'CWP232291' | 0, 0.25, 0.5, 1, 1.5, 2, 4, 8, 24 hours post-dose
  Peak Plasma Concentration (Cmax) of metabolites of 'CWP232291'
AUC as a pharmacokinetic parameter of metabolites of 'CWP232291' | 0, 0.25, 0.5, 1, 1.5, 2, 4, 8, 24 hours post-dose
  Area under the plasma concentration versus time curve (AUC) of metabolites of 'CWP232291'

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- South Korea (3):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Derived] Lee JH, Faderl S, Pagel JM, Jung CW, Yoon SS, Pardanani AD, Becker PS, Lee H, Choi J, Lee K, Kim M, Cortes JE. Phase 1 study of CWP232291 in patients with relapsed or refractory acute myeloid leukemia and myelodysplastic syndrome. Blood Adv. 2020 May 12;4(9):2032-2043. doi: 10.1182/bloodadvances.2019000757. PMID 32396615